CLINICAL TRIAL: NCT03871140
Title: Intelligent Diagnosis of Focal Liver Lesions and Thermal Ablation Zone of Liver Cancer Based on Ultrasound Imaging
Brief Title: Utility of Ultrasound Imaging for Diagnosis of Focal Liver Lesions: A Radiomics Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Prof, Chinese PLA General Hospital
Other Study IDs: 301jrcsk3
Record Dates: First submitted 2018-04-29; First posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2018-04

CONDITIONS: Focal Liver Lesions; Ultrasonics; Intelligent Diagnosis; Ablation; Radiomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: diagnosis — therre is no intervention diagnosis or treatment for patients

SUMMARY:
Ultrasound (US) as first-line imaging technology in detecting focal liver lesions,also plays a crucial role in evaluating image and guiding ablation which is the main treatment for liver lesions. However, the effect of US in diagnosing liver lesions is challenged by several factors including being highly dependent on doctor's experience, low signal-to-noise ratio, low resolution for lesion feature,large error from thermal field evaluation during the process of ablation and so on. Therefore, it is of great significance to construct an intelligent US analysis system depending on the digital information technology. Basing on these problems,the following research will be involved in our project: 1) US database of liver lesions with seamless connection to Picture Archiving and Communication Systems (PACS) will be developed, with the aim to provide standard data for intelligent US analysis. 2) Deep learning model for accurate segmentation, detection and classification of liver lesions on US images will be studied. Then automatic extraction, selection and analysis of liver lesion ultrasound features and the intelligent US diagnosis for liver lesions will be realized. 3) Proposing a clustering model with deep image features, and depicting the similarity measurement of liver cancer, which can be furthered used to link the liver cancer feature to optimal ablation parameters. The intelligent decision-making system for quantifying thermal ablation will be established. 4) Regression algorithm and Generative Adversarial Nets will be developed to extract the image features of liver cancer which will predict risk factors after US-guided thermal ablation.Based on the above researches, it is of great value to establish an intelligent focal liver lesion US diagnosis system involving intelligent diagnosis,personalized ablation strategy and accurate prognosis evaluation, improving the level of accurate diagnosis and treatment of liver lesions.

ELIGIBILITY:
Inclusion Criteria:

1. clear ultrasound imaging of focal liver lesions including malignant liver tumors such as hepatocellular carcinoma, metastatic liver cancer and benigh liver tumors such as hemangioma and focal nodular hyperplasia and so on can be acquired.
2. clear ultrasound imaging of liver tissues backgroud without lesions can be acquired.
3. disease history and pathological diagnosis of the lesions can be acquired.

Exclusion Criteria:

1. patients unsuitable for ultrasound san
2. patients counldn't provide disease history such as hepatitis, alcohol intake and so on
3. patients without pathological results

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with focal liver lesions
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
AUC value | through study completion, an average of 3 year
  Area under the receiver operating characteristic (ROC) curve (AUC）
specificity | through study completion, an average of 3 year
  diagnosis specificity of intelligent ultrasound analysis
sensitivity | through study completion, an average of 3 year
  diagnosis sensitivity of intelligent ultrasound analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Du Z, Fan F, Ma J, Liu J, Yan X, Chen X, Dong Y, Wu J, Ding W, Zhao Q, Wang Y, Zhang G, Yu J, Liang P. Development and validation of an ultrasound-based interpretable machine learning model for the classification of </=3 cm hepatocellular carcinoma: a multicentre retrospective diagnostic study. EClinicalMedicine. 2025 Feb 13;81:103098. doi: 10.1016/j.eclinm.2025.103098. eCollection 2025 Mar. PMID 40034568
- [Derived] Yang Y, Cairang Y, Jiang T, Zhou J, Zhang L, Qi B, Ma S, Tang L, Xu D, Bu L, Bu R, Jing X, Wang H, Zhou Z, Zhao C, Luo B, Liu L, Guo J, Nima Y, Hua G, Wa Z, Zhang Y, Zhou G, Jiang W, Wang C, De Y, Yu X, Cheng Z, Han Z, Liu F, Dou J, Feng H, Wu C, Wang R, Hu J, Yang Q, Luo Y, Wu J, Fan H, Liang P, Yu J. Ultrasound identification of hepatic echinococcosis using a deep convolutional neural network model in China: a retrospective, large-scale, multicentre, diagnostic accuracy study. Lancet Digit Health. 2023 Aug;5(8):e503-e514. doi: 10.1016/S2589-7500(23)00091-2. PMID 37507196